CLINICAL TRIAL: NCT05248594
Title: Real World Use of Emicizumab in Infants and Children Ages 0-3 Years With Hemophilia A
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Genentech, Inc. (Industry); Regional Comprehensive Hemophilia Treatment Center (Mount Sinai) (Unknown); Massachusetts General Comprehensive Hemophilia and Thrombosis Treatment Center (Unknown); Rutgers Robert Wood Johnson Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-13264; ML43506 (Other: Sponsor)
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: HEMLIBRA — Emicizumab (Hemlibra, also known as ACE910 and RO5534262) is a humanized monoclonal modified immunoglobulin G4 (IgG4) antibody with a bispecific antibody structure produced by recombinant DNA technology in Chinese hamster ovary (CHO) cells.
  Other Names: Emicizumab-kxwh

SUMMARY:
Hemophilia A (HA) is a rare congenital bleeding disorder characterized by coagulation factor VIII deficiency. In severe HA, defined as plasma FVIII clotting activity < 1%, bleeding may frequently occur spontaneously, most commonly in joints, leading to painful hemophilic arthropathy and loss of joint function. Patients with moderate or mild hemophilia A, defined as FVIII clotting activity between 1-<5% and 5-40% respectively, are less likely to have spontaneous bleeding however can have significant bleeding with trauma or surgery. Perioperative management by a hematologist who specializes in hemophilia is needed to ensure hemostasis during surgery. Hemophilia is an X-linked recessive disorder affecting 1 in 5000 to 10,000 males.

DETAILED DESCRIPTION:
A questionnaire to elucidate the dosing, frequency and indication for the use of emicizumab in patients with Hemophilia A (mild, moderate or severe) ages 0-3 years has been developed. Data on any pre-, peri and post-surgical practices while on emicizumab is being collected. Pediatricians are being asked if there are plans to introduce factor 8 to children who are already on emicizumab for primary prophylaxis as well as how and when this is planned on being done. The hope is that this data will help inform understanding of current use of emicizumab in infants and young children as a form of primary prophylaxis, especially when venous access has historically been a limiting factor.

This will be a multi-institutional, retrospective review of pediatric patients ages 0 to 36 months of age who are currently receiving and/or have received emicizumab-kxwh as part of their treatment for hemophilia A with or without inhibitors. Participating sites are part of the New England Region (plus New Jersey and New York-Region II) of hemophilia treatment centers. Each institution will be contributing subjects who have been treated or who are currently being treated with emicizumab, from October 4th, 2018 up to the point of IRB approval. Additionally, each institution will determine the best way to identify eligible patients and keep track of patients enrolled in the study. The Children's Hospital at Montefiore will be the coordinating center.

ELIGIBILITY:
Inclusion Criteria: Patients must meet the following criteria for study entry:

* Patients who have been prescribed Emicizumab
* Patients who are 0-36 months of age at the time of starting treatment with Emicizumab
* Diagnosis of congenital mild, moderate or severe hemophilia with or without an inhibitor

Exclusion Criteria:

* Patients with acquired Hemophilia A
* Patients with Hemophilia A and another congenital or acquired bleeding disorder.

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients 0 to 36 months of age, diagnosed with severe, moderate or mild Hemophlia A at the time of initiating treatment with Emicizumab.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
The proportion of patients that are being treated with emicizumab | Within a year.
  The primary outcome will include the proportion of patients that are being treated with emicizumab for primary prophylaxis, as well as identifying breakthrough bleeding while on emicizumab.

SECONDARY OUTCOMES:
Patients who receive additional doses of factor concentrate while on emicizumab | Within a year.
  Data collected will also include proportion of patients who receive additional doses of factor concentrate while on emicizumab for trauma or surgical interventions.

OTHER OUTCOMES:
Patients by demographics (age and race), clinical (severity of hemophilia, inhibitor history) and treatment data | Within a year.
  Additionally, we will characterize the 37+ patients by demographics (age and race), clinical (severity of hemophilia, inhibitor history) and treatment data (indication for emicizumab ie. primary vs secondary prophylaxis.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Davila, MD, Principal Investigator — Children's Hospital at Montefiore
Locations (10):
- United States (10):
  - Connecticut Children's Hemophilia Treatment Center - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale Hemophilia Treatment Center, New Haven, Connecticut
  - Dartmouth Hitchcock Hemophilia Center - Mary Hitchcock Memorial Hospital, Lebanon, New Hampshire
  - Newark Beth Israel, Newark, New Jersey
  - Western NY Blood Care - Research Foundation for SUNY, Buffalo, New York
  - Comprehensive Center for Hemophilia and Coagulation Disorders (Cornell), New York, New York
  - Mary M Gooley Hemophilia Center, Inc., Rochester, New York
  - Northwell Health Hemostasis and Thrombosis Center, Staten Island, New York
  - SUNY Upstate Hemophilia Treatment Center - HTC 058, Syracuse, New York
  - Children's Hospital at Montefiore, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No